CLINICAL TRIAL: NCT03600350
Title: Phase II Trial of a DNA Vaccine Encoding Prostatic Acid Phosphatase (pTVG-HP) and Nivolumab in Patients With Non-Metastatic, PSA-Recurrent Prostate Cancer
Brief Title: pTVG-HP and Nivolumab in Patients With Non-Metastatic PSA-Recurrent Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Bristol-Myers Squibb (Industry); Madison Vaccines Inc. (MVI) (Unknown); AIQ Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW18008; 2018-0418 (Other: IRB Number); A534260 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); NCI-2018-01474 (Registry Identifier: NCI Trial ID); Protocol Version 4/15/2024 (Other: UW Madison)
Record Dates: First submitted 2018-07-11; First posted 2018-07-26 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nivolumab; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Intervention Model Description: Single-arm, single-institution, two-stage phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): * Nivolumab 240 mg IV every two weeks x 6 beginning day 1, then every four weeks x 9 beginning week 12
  * pTVG-HP (100 µg) administered intradermally (i.d.) every two weeks x 6 beginning day 1, then every four weeks x 9 beginning week 12
  * rhGM-CSF (208 µg) administered intradermally (i.d.) every two weeks x 4 beginning week 4, then every four weeks x 9 beginning week 12 NOTE: Only administered to patients for whom serum PSA obtained week 4 > serum PSA obtained at day 1.
  Interventions: Biological: pTVG-HP; Drug: Nivolumab; Drug: GM-CSF

INTERVENTIONS:
Biological: pTVG-HP — Plasmid DNA vaccine encoding Prostatic Acid Phosphatase (PAP)
Drug: Nivolumab — Nivolumab is a human programmed death receptor-1 (PD-1)-blocking antibody indicated for the treatment of patients with multiple different types of cancer.
  Other Names: Opdivo
Drug: GM-CSF — Granulocyte-macrophage colony-stimulating factor (GM-CSF) is a growth factor that supports the survival, clonal expansion and differentiation of hematopoietic progenitor cells including dendritic antigen presenting cells.
  Other Names: Leukine; Sargramostim

SUMMARY:
The purpose of this study is to evaluate the safety of an investigational DNA vaccine, pTVG-HP, a plasmid DNA encoding human prostatic acid phosphatase (PAP), in combination with nivolumab, and the efficacy of this combination in decreasing serum Prostate-Specific Antigen (PSA) in patients with non-metastatic, non-castrate prostate cancer (clinical stage D0/M0).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age with a histologic diagnosis of adenocarcinoma of the prostate
* Patients must have undergone radical prostatectomy
* Patients must have completed local therapy by surgery and any adjuvant/salvage radiation therapy at least 3 months prior to entry, with removal or ablation of all visible disease, including seminal vesical and/or local lymph node involvement.
* Patients must have biochemically recurrent, non-metastatic (by CT and bone scan) clinical stage D0/M0 disease defined by the following:

  * Patients must have evidence of detectable serum PSA with at least 4 serum PSA measurements available, from the same clinical laboratory, at least two weeks apart up to one year, and the final serum PSA value must be > 2.0 ng/mL.
  * PSA doubling time, calculated from most recent 4 serum PSA values (collected up to one year prior to enrollment, at least 2 weeks apart, and all from the same clinical laboratory), must be a positive number (i.e. evidence of PSA rise over time).
  * PSA doubling time will be calculated using the Memorial Sloan-Kettering Cancer Center nomogram (http://www.mskcc.org/applications/nomograms/prostate/PsaDoublingTime.aspx).
  * Patients must not have definitive evidence of metastases as determined by CT of the abdomen/pelvis and bone scintigraphy (bone scan). Note: patients with lesions detectable by highly sensitive methods (e.g. NaF PET imaging or PSMA PET imaging) will be considered eligible as long as these lesions do not meet size criteria on CT imaging (visceral lesions suspicious for metastases or lymph node > 15 mm in short axis) and/or are not independently observed on bone scan
* Patients with a prior history of a second malignancy are eligible provided they have been treated with curative intent and have been free of disease greater than three years. There will be no exclusion for patients with a history of basal cell carcinoma, squamous cell skin cancer, superficial bladder cancer, or other in situ carcinoma that has been adequately treated.
* Patients who are sexually active must use a reliable form of contraception while on study and for 4 weeks after the last immunization.
* ECOG performance score < 2 and life expectancy of at least 12 months.
* Patients must have normal hematologic, renal and liver function as defined by: WBC > 3000/mm3, hematocrit > 30%, platelet count > 100,000/mm3, serum creatinine < 1.5 mg/dl or a calculated creatinine clearance > 60 cc/min, AST or ALT < 3.0x ULN, and serum bilirubin < 2.0 mg/dl(except participants with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL), within 4 weeks prior to first immunization.
* Patients must be informed of the experimental nature of the study and its potential risks and must sign an IRB-approved written informed consent form indicating such an understanding.
* Willingness to provide blood samples for immune studies, per study calendar, up to one year after study, even if off study treatment.

Exclusion Criteria:

* Small cell or other variant prostate cancer histology
* Patients cannot have evidence of immunosuppression or have been treated with immunosuppressive therapy, such as chemotherapy or chronic treatment dose corticosteroids (greater than the equivalent of 10 mg prednisone per day), within 3 months of the first vaccination.
* Seropositive for HIV, hepatitis B (HBV) or hepatitis C (HCV) per patient history due to the immunosuppressive features of these diseases.
* Prior treatment with an LHRH agonist or nonsteroidal antiandrogen, except in the following circumstances: Neoadjuvant/adjuvant androgen deprivation therapy administered with radiation therapy or at the time of prostatectomy is acceptable, provided that there was no evidence of PSA progression while on treatment. In this situation, patients must not have received more than 24 months of androgen deprivation treatment. Other treatment with androgen deprivation therapy is prohibited.
* Serum testosterone at screening < 50 ng/dL.
* Patients must not be concurrently taking other medications or supplements with known hormonal effects, including PC-SPES, megestrol acetate, finasteride, ketoconazole, estradiol, or Saw Palmetto. All other medications with possible anticancer effects must be discussed with the PI prior to study entry.
* Patients previously treated with herbal supplements as described in 5.B.6 or other potential or experimental therapies for prostate cancer must have discontinued these treatments and completed at least a 4 week washout prior to beginning treatment.
* Patients must not have evidence of bone metastases or lymph node involvement as determined by bone scan or CT scan of the abdomen and pelvis within 4 weeks of study registration. Note: Advanced imaging modalities (such as NaF-PET/CT, choline PET/CT, fluciclovine, or PSMA PET scans) will NOT be used to determine evidence of metastases for eligibility purposes or for defining disease progression.
* Patients must not have been treated with a prior DNA vaccine therapy for prostate cancer.
* Patients must not have known psychological or sociological conditions, addictive disorders or family problems, which would preclude compliance with the protocol.
* Patients must not have known allergic reactions to GM-CSF.
* Patients with unstable or severe intercurrent medical conditions or laboratory abnormalities that would impart, in the judgment of the PI, excess risk associated with study participation or study agent administration.
* Patients cannot have concurrent enrollment on other phase I, II, or III investigational therapeutic treatment studies.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Emamekhoo, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Derived] McNeel DG, Emamekhoo H, Eickhoff JC, Kyriakopoulos CE, Wargowski E, Tonelli TP, Johnson LE, Liu G. Phase 2 trial of a DNA vaccine (pTVG-HP) and nivolumab in patients with castration-sensitive non-metastatic (M0) prostate cancer. J Immunother Cancer. 2023 Dec 14;11(12):e008067. doi: 10.1136/jitc-2023-008067. PMID 38101860
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from September 2018 to December 2021.
Groups:
- Treatment Group: * Nivolumab 240 mg IV every two weeks x 6 beginning day 1, then every four weeks x 9 beginning week 12
  * pTVG-HP (100 µg) administered intradermally (i.d.) every two weeks x 6 beginning day 1, then every four weeks x 9 beginning week 12
  * rhGM-CSF (208 µg) administered intradermally (i.d.) every two weeks x 4 beginning week 4, then every four weeks x 9 beginning week 12 NOTE: Only administered to patients for whom serum PSA obtained week 4 > serum PSA obtained at day 1.
  pTVG-HP: Plasmid DNA vaccine encoding Prostatic Acid Phosphatase (PAP)
  Nivolumab: Nivolumab is a human programmed death receptor-1 (PD-1)-blocking antibody indicated for the treatment of patients with multiple different types of cancer.
  GM-CSF: Granulocyte-macrophage colony-stimulating factor (GM-CSF) is a growth factor that supports the survival, clonal expansion and differentiation of hematopoietic progenitor cells including dendritic antigen presenting cells.
Period: Overall Study
Arm/Group | Treatment Group
Started | 19
On Treatment | 19
Off Treatment | 19
Completed | 0
Not Completed | 19
Not completed — Death | 1
Not completed — On Follow Up | 18

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
Age, Customized [Count of Participants; unit: Participants]
  60-69 years | 10
  70-79 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events Grade 3 or Higher
Description: Subjects will be evaluated at each visit by a review of systems based on the most recent version of the NCI common toxicity criteria. Safety and Tolerability of this intervention is defined as following: a toxicity rate p0 of at most 15% of Grade ≥ 3 toxicity events (CTCAE v.4.0) will be considered as acceptable while a toxicity rate p1=35% or more will be considered as unacceptably high. See Adverse Events Section for full summary of data.
Time Frame: up to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
Participants | 4

2. Primary Outcome: Prostate-Specific Antigen (PSA) Complete Response (CR) Rate
Description: A PSA CR will be defined as the percentage of participants with a serum PSA <0.2 ng/mL and confirmatory PSA <0.2 ng/mL at least 4 weeks later, as per Prostate Cancer Working Group 2 (PCWG2) recommendations. To qualify as a PSA CR, there must be no evidence of radiographic progression.
Time Frame: up to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
Participants | 0

3. Secondary Outcome: Metastasis-free Survival Rate
Description: The 5-year metastasis-free survival will be determined by investigator review of radiographic studies (CT/MRI and bone scintigraphy) performed 5 years after study initiation in subjects who have not already met criteria for radiographic progression.
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Median Radiographic Progression-free Survival
Description: All participants will undergo radiographic imaging prior to treatment and at 6-month intervals (or as clinically required). The appearance of lesions consistent with metastatic disease will be used to define radiographic progression.
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: PSA Doubling Time
Description: Post-treatment doubling time will be calculated from: 1) All PSA values obtained from the same clinical laboratory using the same PSA assay beginning with the PSA value at day 1 (week 0) and continuing until the end-of study (or month 24) value (PSADT 0-24). 2) All PSA values obtained from the same clinical laboratory using the same PSA assay beginning with the PSA value at day 85 (month 3) to the day 253 (month 9) value (PSADT 3-9).
Time Frame: Up to 2 years
Reporting Status: Not Posted

6. Secondary Outcome: PSA Response Rate (</= 50% of Baseline)
Description: The percentage of participants with PSA values less than or equal to their baseline value after 2 year.
Time Frame: Up to 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Number of Participants Receiving GM-CSF as an Adjuvant After Week 4
Description: GM-CSF is used as an adjuvant if the PSA at week 4 is higher than baseline.
Time Frame: up to week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
Participants | 14

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 1/19
Serious Adverse Events (participants affected / at risk) | 5/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=19)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=19)
Fatigue (General disorders) | 11 (15)
Chills (General disorders) | 6 (10)
Injection site reaction (General disorders) | 4 (8)
Non-cardiac chest pain (General disorders) | 3 (3)
Fever (General disorders) | 2 (5)
Pain (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (10)
Abdominal pain (Gastrointestinal disorders) | 4 (8)
Bloating (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Serum amylase increased (Investigations) | 4 (5)
Creatinine increased (Investigations) | 3 (3)
Lipase increased (Investigations) | 2 (8)
Lymphocyte count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 3 (5)
Tremor (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (9)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 2 (3)
Lung infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hypertension (Vascular disorders) | 5 (9)
Hot flashes (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (5)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (7)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT03600350/Prot_SAP_000.pdf